CLINICAL TRIAL: NCT04160468
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of a Single Dose of Exebacase in Patients Receiving Standard-of-Care Antibiotics for the Treatment of Staphylococcus Aureus Bloodstream Infections (Bacteremia), Including Right-Sided Infective Endocarditis
Brief Title: Direct Lysis of Staph Aureus Resistant Pathogen Trial of Exebacase
Acronym: DISRUPT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The independent DSMB recommended that the study be stopped for futility following interim efficacy analysis.
Sponsor: ContraFect (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF-301-105
Record Dates: First submitted 2019-11-07; First posted 2019-11-13 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Staphylococcus Aureus Bacteremia; Staphylococcus Aureus Endocarditis
Keywords: S. aureus bloodstream infection; S. aureus bacteremia; S. aureus right-sided infective endocarditis
MeSH Terms: interventions — exebacase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Exebacase (Experimental)
  Interventions: Drug: Exebacase
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exebacase — Participants will receive a single IV infusion of exebacase in addition to SoCA selected by the investigator. Participants with normal renal function or mild renal impairment will be administered a dose of 18 mg; participants with moderate or severe renal impairment will be administered a dose of 12 mg of exebacase; participants with end-stage renal disease, including those on hemodialysis, will be administered a dose of 8 mg of exebacase.
  Arms: Exebacase
Drug: Placebo — Participants will receive a single IV infusion of placebo in addition to SoCA selected by the investigator.
  Arms: Placebo

SUMMARY:
The purpose of this superiority study is to evaluate the efficacy and safety of exebacase in addition to standard of care antibiotics (SoCA) compared with SoCA alone for the treatment of patients with Staphylococcus aureus (S. aureus) bloodstream infections (BSI), including right-sided infective endocarditis (IE). Patients will be randomized to receive a single intravenous dose of exebacase or placebo. Patients will receive SoCA selected by the investigators based on the protocol.

Exebacase, a direct lytic agent, is an entirely new treatment modality against S. aureus. Exebacase is a recombinantly-produced, purified cell wall hydrolase enzyme that results in rapid bacteriolysis, potent biofilm eradication, synergy with antibiotics, low propensity for resistance, and the potential to suppress antibiotic resistance when used together with antibiotics. Exebacase represents a first-in-field, first-in-class treatment with the potential to improve clinical outcome when used in addition to SoCA to treat S. aureus BSI including IE.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 12 years or older
* Blood culture positive for S. aureus
* At least two signs or symptoms attributable to S. aureus BSI/IE
* Known or suspected complicated S. aureus BSI and/or right-sided IE based on Modified Duke Criteria
* Not pregnant or breastfeeding and not of reproductive potential or agrees to remain abstinent or use contraception if of reproductive potential

Exclusion Criteria:

* Previously received exebacase
* Known or suspected left-sided IE
* Treatment with effective systemic anti-staphylococcal antibiotic for more than 72 hours within 7 days before randomization
* Presence of prosthetic valve or cardiac valve support ring, or presence of known or suspected infected hardware (orthopedic), prosthetic joint, or cardiac device
* Known polymicrobial BSI, or known ongoing systemic infection caused by other bacterial and/or fungal pathogen(s), and/or known to have coronavirus disease 2019 (COVID-19)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (50):
  - Cf 301-105, Birmingham, Alabama
  - CF-301-105 Study Site, Orange, California
  - Cf 301-105, Sacramento, California
  - Cf 301-105, San Diego, California
  - CF-301-105 Investigator Site, Sylmar, California
  - Cf 301-105, Torrance, California
  - CF-301-105 Study Site, Hartford, Connecticut
  - Cf 301-105, New Haven, Connecticut
  - Cf 301-105, Washington D.C., District of Columbia
  - Cf 301-105, Gainesville, Florida
  - Cf 301-105, Atlanta, Georgia
  - Cf 301-105, Augusta, Georgia
  - Cf 301-105, Decatur, Georgia
  - CF-301-105 Study Site, Idaho Falls, Idaho
  - CF-301-105 Investigator Site, Chicago, Illinois
  - Cf 301-105, Glenview, Illinois
  - Cf 301-105, Highland Park, Illinois
  - Cf 301-105, Maywood, Illinois
  - Cf 301-105, Fort Wayne, Indiana
  - Cf 301-105, Kansas City, Kansas
  - Cf 301-105, Baltimore, Maryland
  - CF 301-105 Study Site, Boston, Massachusetts
  - CF-301-105 Study Site, Burlington, Massachusetts
  - Cf 301-105, Worcester, Massachusetts
  - Cf 301-105, Detroit, Michigan
  - Cf 301-105, Royal Oak, Michigan
  - Cf 301-105, Rochester, Minnesota
  - CF-301-105 Study Site, Columbia, Missouri
  - Cf 301-105, St Louis, Missouri
  - CF-301-105 Study Site, Butte, Montana
  - Cf 301-105, Omaha, Nebraska
  - Cf 301-105, Neptune City, New Jersey
  - Cf 301-105, Newark, New Jersey
  - Cf 301-105, New York, New York
  - Cf 301-105, Valhalla, New York
  - Cf 301-105, Chapel Hill, North Carolina
  - Cf 301-105, Charlotte, North Carolina
  - Cf 301-105, Durham, North Carolina
  - CF-301-105 Study Site, Greenville, North Carolina
  - CF-301-105 Study Site, Columbus, Ohio
  - Cf 301-105, Toledo, Ohio
  - Cf 301-105, Allentown, Pennsylvania
  - Cf 301-105, Philadelphia, Pennsylvania
  - CF 301-105 Investigator Site, West Reading, Pennsylvania
  - Cf 301-105, Memphis, Tennessee
  - Cf 301-105, Nashville, Tennessee
  - Cf 301-105, Houston, Texas
  - CF-301-105 Study Site, Salt Lake City, Utah
  - Cf 301-105, Burlington, Vermont
  - Cf 301-105, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Fowler VG Jr, Das AF, Lipka-Diamond J, Ambler JE, Schuch R, Pomerantz R, Cassino C, Jauregui-Peredo L, Moran GJ, Rupp ME, Lachiewicz AM, Kuti JL, Wise RA, Kaye KS, Zervos MJ, Nichols WG. Exebacase in Addition to Standard-of-Care Antibiotics for Staphylococcus aureus Bloodstream Infections and Right-Sided Infective Endocarditis: A Phase 3, Superiority-Design, Placebo-Controlled, Randomized Clinical Trial (DISRUPT). Clin Infect Dis. 2024 Jun 14;78(6):1473-1481. doi: 10.1093/cid/ciae043. PMID 38297916
- [Derived] Traczewski MM, Ambler JE, Schuch R. Determination of MIC Quality Control Parameters for Exebacase, a Novel Lysin with Antistaphylococcal Activity. J Clin Microbiol. 2021 Jun 18;59(7):e0311720. doi: 10.1128/JCM.03117-20. Epub 2021 Jun 18. PMID 33910968

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 348 patients were planned, and 259 patients were randomized at the time the study was stopped for futility.
Groups:
- Exebacase + SoCA: Participants received a single IV infusion of exebacase in addition to standard-of-care antibiotics (SoCA) selected by the investigator.
- SoCA Alone: Participants received a single IV infusion of placebo in addition to standard-of-care antibiotics (SoCA) selected by the investigator.
Period: Overall Study
Arm/Group | Exebacase + SoCA | SoCA Alone
Started | 173 | 86
Completed | 142 | 81
Not Completed | 31 | 5
Not completed — Lost to Follow-up | 19 | 4
Not completed — Randomized but not dosed | 6 | 0
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Participant unable/unwilling to adhere to protocol | 1 | 0
Not completed — Participant incarcerated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Microbiological intent-to-treat (mITT) analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Exebacase + SoCA | SoCA Alone | Total
Number analyzed (Participants) | 165 | 85 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 119 | 63 | 182
  >=65 years | 44 | 22 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 48 | 158
  Male | 55 | 37 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 10 | 30
  Not Hispanic or Latino | 138 | 75 | 213
  Unknown or Not Reported | 7 | 0 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 28 | 16 | 44
  White | 118 | 65 | 183
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 1 | 12
Region of Enrollment [Number; unit: participants]
  United States | 165 | 85 | 250
Final Adjudicated Diagnosis [Count of Participants; unit: Participants] — Patients with S. aureus right-sided infective endocarditis, complicated bloodstream infection, or risk factors for complicated bloodstream infection were eligible. Patients with left-sided infective endocarditis or uncomplicated bloodstream infections were excluded from the study based on the investigator's assessment. The diagnosis of complicated bloodstream infection, uncomplicated bloodstream infection, right-sided infective endocarditis, and left-sided infective endocarditis reported on this table are based on the Adjudication Committee's determination of final adjudicated diagnosis.
  Participants
    Complicated bloodstream infection | 127 | 63 | 190
    Uncomplicated bloodstream infection | 11 | 9 | 20
    Right-sided infective endocarditis | 22 | 10 | 32
    Left-sided infective endocarditis | 4 | 3 | 7
    Right- and left-sided infective endocarditis | 1 | 0 | 1
Methicillin-resistant S. aureus (MRSA) and methicillin-susceptible S. aureus (MSSA) [Count of Participants; unit: Participants]
  MRSA | 64 | 33 | 97
  MSSA | 101 | 52 | 153

OUTCOME MEASURES:

1. Primary Outcome: Clinical Responder Rate at Day 14 in the MRSA Population in the Microbiological Intent-to-treat (mITT) Analysis Set
Description: Clinical outcome of responder was defined as survival with resolution or 2-grade improvement of attributable signs and symptoms and negative blood cultures by Day 14, and without new signs or symptoms, new metastatic foci or septic emboli, or change in antibiotics due to lack of response.
Time Frame: Day 14
Population: MRSA population in the mITT analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Exebacase + SoCA | SoCA Alone
Number analyzed (Participants) | 64 | 33
Participants
  Responder | 32 | 20
  Failure | 30 | 13
  Indeterminate | 2 | 0
Statistical Analysis 1: Comparison: Exebacase + SoCA vs SoCA Alone; Test type: Superiority; p = 0.392, Fisher Exact; Risk Difference (RD) = -10.6, 95% CI 2-sided [-33.6 to 12.4]

2. Primary Outcome: Treatment-emergent Adverse Events (TEAEs) Through Day 60
Description: Number and percentage of patients with treatment-emergent adverse events (TEAEs)
Time Frame: Through Day 60
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Exebacase + SoCA | SoCA Alone
Number analyzed (Participants) | 165 | 85
Participants | 142 | 72

ADVERSE EVENTS:
Time Frame: Through the Day 60 visit
Description: All adverse events (AEs) and serious adverse events (SAEs) were collected from the time of consent through the Day 60 visit. Treatment emergent AEs, defined as an AE that occurred during or after study drug administration through the Day 60 visit (Day 60 ±7 days), are presented in the overall population in the safety analysis set.
Arm/Group | Exebacase + SoCA | SoCA Alone
All-Cause Mortality (participants affected / at risk) | 27/165 | 14/85
Serious Adverse Events (participants affected / at risk) | 71/165 | 34/85
Other Adverse Events (participants affected / at risk) | 72/165 | 41/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exebacase + SoCA (N=165) | SoCA Alone (N=85)
Staphylococcal bacteremia (Infections and infestations) | 3 | 1
Osteomyelitis (Infections and infestations) | 2 | 2
Septic shock (Infections and infestations) | 2 | 2
Pneumonia (Infections and infestations) | 1 | 3
Endocarditis (Infections and infestations) | 1 | 2
Clostridium difficile infection (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
Bone abscess (Infections and infestations) | 1 | 0
Cavernous sinus thrombosis (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Pharyngeal abscess (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 2
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Candida sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 1 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 2
End stage renal disease (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Gastrointestinal hemorrage (Gastrointestinal disorders) | 3 | 0
Intestinal angioedema (Gastrointestinal disorders) | 1 | 0
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Peritoneal hematoma (Gastrointestinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 0
Shock (Vascular disorders) | 2 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0
Acute disseminated encephalomyelitis (Nervous system disorders) | 1 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Subarachnoid hemorrhage (Nervous system disorders) | 1 | 0
Ischemic stroke (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 0 | 1
Death NOS (not otherwise specified) (General disorders) | 3 | 3
Death (General disorders) | 2 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Ischemic hepatitis (Hepatobiliary disorders) | 2 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Chronic hepatic failure (Hepatobiliary disorders) | 0 | 1
Wound dehiscense (Injury, poisoning and procedural complications) | 2 | 0
Heart injury (Injury, poisoning and procedural complications) | 1 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 2
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Drug abuse (Psychiatric disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Patient dissatisfaction with treatment (Social circumstances) | 1 | 1
Social stay hospitalization (Social circumstances) | 1 | 0
Mixed deafness (Ear and labyrinth disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Device dislocation (Product Issues) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exebacase + SoCA (N=165) | SoCA Alone (N=85)
Pneumonia (Infections and infestations) | 5 | 6
Urinary tract infection (Infections and infestations) | 3 | 5
Constipation (Gastrointestinal disorders) | 13 | 11
Diarrhea (Gastrointestinal disorders) | 12 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Anemia (Blood and lymphatic system disorders) | 12 | 8
Hypotension (Vascular disorders) | 13 | 9
Deep vein thrombosis (Vascular disorders) | 5 | 5
Acute kidney injury (Renal and urinary disorders) | 16 | 8
Urinary retention (Renal and urinary disorders) | 7 | 6
Rash (Skin and subcutaneous tissue disorders) | 10 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT04160468/Prot_SAP_000.pdf